CLINICAL TRIAL: NCT02884674
Title: Stimulation magnétique transcrânienne répétitive Dans le Traitement Des Troubles Obsessionnels Compulsifs
Brief Title: Repetitive Transcranial Magnetic Stimulation in Obsessive Compulsive Disorder
Acronym: MAGTOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38RC14.156; 2014-A00668-39 (Other: ID RCB)
Record Dates: First submitted 2015-01-08; First posted 2016-08-31 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active Transcranial Magnetic Stimulation (Active Comparator): Active Transcranial Magnetic Stimulation (TMS) targeting the right frontal inferior gyrus, 2 sessions per day, each session 5min30 day, during 10 consecutive days, Using theta burst stimulation and using Transcranial Magnetic Stimulation navigator and robot
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Placebo (Placebo Comparator): Placebo comparator, using non active magnetic coil, targeting the right frontal inferior gyrus, 2 sessions per day, each session 5min30 day, during 10 consecutive days, using theta burst stimulation and using Transcranial Magnetic Stimulation navigator and robot
  Interventions: Device: Placebo Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation — modulation of the electrical activity of the right inferior frontal gyrus cortex in order to reduce Obsessive Compulsive Disorders symptoms by Active Transcranial Magnetic Stimulation (TMS) targeting the right frontal inferior gyrus, 2 sessions per day, each session 5min30 day, during 10 consecutive days, using theta burst stimulation and using a TMS neuronavigated robot
  Arms: active Transcranial Magnetic Stimulation
Device: Placebo Repetitive Transcranial Magnetic Stimulation — Sham rTMS will be delivered using non active magnetic coil, targeting the right frontal inferior gyrus, 2 sessions per day, each session 5min30 day, during 10 consecutive days, using TMS neuronavigated robot. A subjective sensation will be obtained via frontal dermic electrical stimulation.
  Arms: Placebo

SUMMARY:
Evaluate the therapeutic effect of a functional Magnetic Resonance Imaging (fMRI)-guided and robotized neuronavigated theta burst Transcranial Magnetic Stimulation (TMS) targeting right inferior frontal region in resistant obsessive compulsive disorder (OCD) in a double-blind, randomized, placebo-controlled, monocentric study.

DETAILED DESCRIPTION:
This study evaluates the therapeutic effect of a fMRI-guided and robotized neuronavigated theta burst Transcranial Magnetic Stimulation (TMS) targeting right inferior frontal region in resistant obsessive compulsive disorder (OCD) in a double-blind, randomized, placebo-controlled, monocentric study. The study will also assess the interest of some clinical, neuropsychological, neuroimaging, electrophysiological variables in response prediction, besides physiopathological information.

There is an increasing interest in developping treatments for resistant OCD, which are not responding to the conventional treatment, represented by pharmacotherapy associated to cognitive behavioral therapy. Repetitive TMS represents a promising non invasive brain stimulation approach, but efficacy, best available brain target, optimal responder profile and stimulation parameters need to be further documented.

In this study, the included patients will be randomly assigned to an active (theta burst TMS) or sham-placebo treatment group. TMS will be added to their stable pharmacotherapy. The brain target, the right inferior frontal region, involved in the inhibition control brain network, will be defined in a personalized manner via a fMRI paradigm for each patient. TMS will be delivered daily for 2 successive weeks. Measures of different clinical, neuropsychological , electrophysiological (cortical excitability) variables will be performed at baseline, as well as at the end of the TMS course, and 1 week after. Other assessments are planned at 3 and 6 months, in order to highlight the evolution of the potential benefit.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subjects with Obsessive Compulsive Disorders (OCD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM IV-TR) criteria and validated by an experimented clinician following instruments like SCID (Structured Clinical Interview for DSM IV) or MINI (Mini-International Neuropsychiatric Interview)
* with or without associated tics ("Gilles de la Tourette" Syndrome)
* Age > 18 years old
* Y-BOCS score > 20 and CGI (Clinical Global Impression Scale) score ≥ 4
* Resistant patients to standard treatments - where treatment resistance is defined by partial but insufficient response (Global Assessment of Functioning score GAF score < 60 and/or reduction of Yale Brown Obsessions and Compulsion Scale score < 35%) or lack of response to previous well conducted treatment including:

  * pharmacotherapy : optimal tolerated dose and adequate duration (> 12 weeks) of at least 2 Serotonin Reuptake Inhibitors (selective serotonin reuptake inhibitors, clomipramine), and one augmentation strategy (adjunction of an antipsychotic - such as risperidone or olanzapine or aripiprazole - or lithium or buspirone) ;
  * psychotherapy (at least 6 months of cognitive and behavioral therapy)

Exclusion Criteria:

* other primary diagnosis than OCD (comorbid tics and depression are tolerated)
* comorbid diagnosis of schizophrenia/ psychotic disorder, bipolar disorder, substance abuse or dependance
* medical condition involving cognitive decline and affecting brain structures such as Parkinson disease, dementia, multiple sclerosis, HIV (human immunodeficiency virus) infection, lupus etc.
* Magnetic Resonance Imaging exclusion criteria (ferromagnetic implants etc)
* common TMS exclusion criteria (neurological condition with an increased risk of seizure, cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, intracranial implants (e.g. cochlear implants, electrodes, aneurysm clips, stimulators... ) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed will be excluded
* Current use of any investigational drug
* pregnancy / breast feeding patients
* visual or auditive important deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-11 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the score at the Yale - Brown Obsessive and Compulsive Scale | at baseline and at day 21
  Evaluation of Obsessive Compulsive Disorder symptoms using the Yale - Brown Obsessive and Compulsive Scale, at day 21, corresponding to 7 days after the end of the TMS cure, compared to baseline.

SECONDARY OUTCOMES:
Score of Montgomery and Asberg Depression Rating Scale, as a Measure of effects on Mood (depression) | At baseline, at day 21, day 90, day 180
  Evaluation of Mood using Montgomery Asberg Depression Rating Scale
Score of Young Mania Rating Scale, as a Measure of effects on Mood (hyperthymia) | At baseline, at day 21, day 90, day 180
  Evaluation of Mood using Young Mania Rating Scale
Score of Multidimensional Assessment of Thymic States Scale as a Measure of effects on Emotional Reactivity | At baseline, at day 21, day 90, day 180
  Evaluation of Emotional Reactivity using Multidimensional Assessment of Thymic States Scale
Number of patients with Side effects as a measure of Safety and Tolerability | for each session of Transcranial Magnetic Stimulation, at day 15, day 21, day 90, day 180
  collection of the side effects of the Transcranial Magnetic Stimulation, after each session, during the entire TMS cure
Inferior Frontal Region Activity (percentage of the BOLD signal change (parameter estimates beta) | at baseline (day 0)
  Performing a functional Magnetic Resonance Imaging, looking for biomarkers of response to the TMS cure.
  Especially studying the right inferior cortex activation in functional Magnetic Resonance Imaging using a Signal Stop Task.
Fractional Anisotropy (FA), mean and radial diffusivity (MD, RD), tracti integrity of the inhibition network, | at day 0 (baseline)
  looking for anatomical biomarkers of response, or anatomical differences between the subjects on the inhibition network using Diffusing Tensor Imaging data
Yale - Brown Obsessive and Compulsion Scale score after the TMS treatment as an evaluation of the persistence of the clinical benefit | day 15, day 90 and day 180 after the inclusion.
  The Yale - Brown Obsessive and Compulsion Scale will also be performed at day 15, day 90 and day 180 after the inclusion in order to assess the kinetics of clinical changes in Obsessive Compulsive symptoms after the TMS cure.
Cortical Excitability | baseline - day 15 - day 21 - day 90 - day 180
  assessing a new biomarker linked to OCD and monitoring its evolution with the TMS cure, testing its predictive value for the clinical response
Evaluation of Impulsivity using specific scales | At baseline, at day 21, day 90, day 180
  Evaluation of impulsivity using UPPS (Urgency, Premeditation, and Sensation Seeking) Impulsive Behavior Scale.
Evaluation of the Clinical global State | at baseline, day 15, day 21, day 90, day 180
  Using Clinical Global Impression scale we will assess the evolution of the clinical global status
type of side effects (pain, paresthesia, other) as a measure of Safety and Tolerability | for each session of Transcranial Magnetic Stimulation, at day 15, day 21, day 90, day 180
  collection of the side effects of the Transcranial Magnetic Stimulation, after each session, during the entire TMS cure

CONTACTS AND LOCATIONS:
Overall Officials: Mircea POLOSAN, Professor, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- CHU de Grenoble - Pavillon Dominique Villars, Grenoble, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Heyman I, Mataix-Cols D, Fineberg NA. Obsessive-compulsive disorder. BMJ. 2006 Aug 26;333(7565):424-9. doi: 10.1136/bmj.333.7565.424. No abstract available. PMID 16931840
- [Background] Denys D. Pharmacotherapy of obsessive-compulsive disorder and obsessive-compulsive spectrum disorders. Psychiatr Clin North Am. 2006 Jun;29(2):553-84, xi. doi: 10.1016/j.psc.2006.02.013. PMID 16650723
- [Background] Barker AT, Jalinous R, Freeston IL. Non-invasive magnetic stimulation of human motor cortex. Lancet. 1985 May 11;1(8437):1106-7. doi: 10.1016/s0140-6736(85)92413-4. No abstract available. PMID 2860322
- [Background] Baxter LR Jr, Phelps ME, Mazziotta JC, Guze BH, Schwartz JM, Selin CE. Local cerebral glucose metabolic rates in obsessive-compulsive disorder. A comparison with rates in unipolar depression and in normal controls. Arch Gen Psychiatry. 1987 Mar;44(3):211-8. doi: 10.1001/archpsyc.1987.01800150017003. PMID 3493749
- [Background] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Di Lazzaro V, Pilato F, Dileone M, Profice P, Oliviero A, Mazzone P, Insola A, Ranieri F, Meglio M, Tonali PA, Rothwell JC. The physiological basis of the effects of intermittent theta burst stimulation of the human motor cortex. J Physiol. 2008 Aug 15;586(16):3871-9. doi: 10.1113/jphysiol.2008.152736. Epub 2008 Jun 19. PMID 18566003
- [Background] Prasko J, Paskova B, Zalesky R, Novak T, Kopecek M, Bares M, Horacek J. The effect of repetitive transcranial magnetic stimulation (rTMS) on symptoms in obsessive compulsive disorder. A randomized, double blind, sham controlled study. Neuro Endocrinol Lett. 2006 Jun;27(3):327-32. PMID 16816829
- [Background] Sarkhel S, Sinha VK, Praharaj SK. Adjunctive high-frequency right prefrontal repetitive transcranial magnetic stimulation (rTMS) was not effective in obsessive-compulsive disorder but improved secondary depression. J Anxiety Disord. 2010 Jun;24(5):535-9. doi: 10.1016/j.janxdis.2010.03.011. Epub 2010 Mar 29. PMID 20392594
- [Background] Sack AT, Cohen Kadosh R, Schuhmann T, Moerel M, Walsh V, Goebel R. Optimizing functional accuracy of TMS in cognitive studies: a comparison of methods. J Cogn Neurosci. 2009 Feb;21(2):207-21. doi: 10.1162/jocn.2009.21126. PMID 18823235
- [Background] Sachdev PS, McBride R, Loo CK, Mitchell PB, Malhi GS, Croker VM. Right versus left prefrontal transcranial magnetic stimulation for obsessive-compulsive disorder: a preliminary investigation. J Clin Psychiatry. 2001 Dec;62(12):981-4. doi: 10.4088/jcp.v62n1211. PMID 11780880
- [Background] Wu CC, Tsai CH, Lu MK, Chen CM, Shen WC, Su KP. Theta-burst repetitive transcranial magnetic stimulation for treatment-resistant obsessive-compulsive disorder with concomitant depression. J Clin Psychiatry. 2010 Apr;71(4):504-6. doi: 10.4088/JCP.09l05426blu. No abstract available. PMID 20409448
- [Background] Aron AR, Fletcher PC, Bullmore ET, Sahakian BJ, Robbins TW. Stop-signal inhibition disrupted by damage to right inferior frontal gyrus in humans. Nat Neurosci. 2003 Feb;6(2):115-6. doi: 10.1038/nn1003. No abstract available. PMID 12536210
- [Background] Chambers CD, Bellgrove MA, Stokes MG, Henderson TR, Garavan H, Robertson IH, Morris AP, Mattingley JB. Executive "brake failure" following deactivation of human frontal lobe. J Cogn Neurosci. 2006 Mar;18(3):444-55. doi: 10.1162/089892906775990606. PMID 16513008
- [Background] Verbruggen F, Aron AR, Stevens MA, Chambers CD. Theta burst stimulation dissociates attention and action updating in human inferior frontal cortex. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13966-71. doi: 10.1073/pnas.1001957107. Epub 2010 Jul 14. PMID 20631303
- [Background] Duncan J, Owen AM. Common regions of the human frontal lobe recruited by diverse cognitive demands. Trends Neurosci. 2000 Oct;23(10):475-83. doi: 10.1016/s0166-2236(00)01633-7. PMID 11006464
- [Background] Verbruggen F, Schneider DW, Logan GD. How to stop and change a response: the role of goal activation in multitasking. J Exp Psychol Hum Percept Perform. 2008 Oct;34(5):1212-28. doi: 10.1037/0096-1523.34.5.1212. PMID 18823206
- [Background] Boucher L, Palmeri TJ, Logan GD, Schall JD. Inhibitory control in mind and brain: an interactive race model of countermanding saccades. Psychol Rev. 2007 Apr;114(2):376-97. doi: 10.1037/0033-295X.114.2.376. PMID 17500631
- [Background] Chambers CD, Bellgrove MA, Gould IC, English T, Garavan H, McNaught E, Kamke M, Mattingley JB. Dissociable mechanisms of cognitive control in prefrontal and premotor cortex. J Neurophysiol. 2007 Dec;98(6):3638-47. doi: 10.1152/jn.00685.2007. Epub 2007 Oct 17. PMID 17942624
- [Background] Aron AR, Behrens TE, Smith S, Frank MJ, Poldrack RA. Triangulating a cognitive control network using diffusion-weighted magnetic resonance imaging (MRI) and functional MRI. J Neurosci. 2007 Apr 4;27(14):3743-52. doi: 10.1523/JNEUROSCI.0519-07.2007. PMID 17409238
- [Background] Swann N, Tandon N, Canolty R, Ellmore TM, McEvoy LK, Dreyer S, DiSano M, Aron AR. Intracranial EEG reveals a time- and frequency-specific role for the right inferior frontal gyrus and primary motor cortex in stopping initiated responses. J Neurosci. 2009 Oct 7;29(40):12675-85. doi: 10.1523/JNEUROSCI.3359-09.2009. PMID 19812342
- [Background] Hampshire A, Chamberlain SR, Monti MM, Duncan J, Owen AM. The role of the right inferior frontal gyrus: inhibition and attentional control. Neuroimage. 2010 Apr 15;50(3):1313-9. doi: 10.1016/j.neuroimage.2009.12.109. Epub 2010 Jan 4. PMID 20056157
- [Background] Chikazoe J, Jimura K, Asari T, Yamashita K, Morimoto H, Hirose S, Miyashita Y, Konishi S. Functional dissociation in right inferior frontal cortex during performance of go/no-go task. Cereb Cortex. 2009 Jan;19(1):146-52. doi: 10.1093/cercor/bhn065. Epub 2008 Apr 28. PMID 18445602
- [Background] Luders H, Lesser RP, Dinner DS, Morris HH, Wyllie E, Godoy J. Localization of cortical function: new information from extraoperative monitoring of patients with epilepsy. Epilepsia. 1988;29 Suppl 2:S56-65. doi: 10.1111/j.1528-1157.1988.tb05799.x. PMID 3168959
- [Background] Johansen-Berg H, Behrens TE, Robson MD, Drobnjak I, Rushworth MF, Brady JM, Smith SM, Higham DJ, Matthews PM. Changes in connectivity profiles define functionally distinct regions in human medial frontal cortex. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13335-40. doi: 10.1073/pnas.0403743101. Epub 2004 Aug 30. PMID 15340158
- [Background] Marsh R, Horga G, Parashar N, Wang Z, Peterson BS, Simpson HB. Altered activation in fronto-striatal circuits during sequential processing of conflict in unmedicated adults with obsessive-compulsive disorder. Biol Psychiatry. 2014 Apr 15;75(8):615-22. doi: 10.1016/j.biopsych.2013.02.004. Epub 2013 Mar 13. PMID 23489416
- [Background] de Wit SJ, de Vries FE, van der Werf YD, Cath DC, Heslenfeld DJ, Veltman EM, van Balkom AJ, Veltman DJ, van den Heuvel OA. Presupplementary motor area hyperactivity during response inhibition: a candidate endophenotype of obsessive-compulsive disorder. Am J Psychiatry. 2012 Oct;169(10):1100-8. doi: 10.1176/appi.ajp.2012.12010073. PMID 23032388
- [Background] Stein DJ, Goodman WK, Rauch SL. The cognitive-affective neuroscience of obsessive-compulsive disorder. Curr Psychiatry Rep. 2000 Aug;2(4):341-6. doi: 10.1007/s11920-000-0079-2. PMID 11122979
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Stokes MG, Chambers CD, Gould IC, Henderson TR, Janko NE, Allen NB, Mattingley JB. Simple metric for scaling motor threshold based on scalp-cortex distance: application to studies using transcranial magnetic stimulation. J Neurophysiol. 2005 Dec;94(6):4520-7. doi: 10.1152/jn.00067.2005. Epub 2005 Aug 31. PMID 16135552
- [Background] Stokes MG, Chambers CD, Gould IC, English T, McNaught E, McDonald O, Mattingley JB. Distance-adjusted motor threshold for transcranial magnetic stimulation. Clin Neurophysiol. 2007 Jul;118(7):1617-25. doi: 10.1016/j.clinph.2007.04.004. Epub 2007 May 23. PMID 17524764
- [Background] Buch ER, Mars RB, Boorman ED, Rushworth MF. A network centered on ventral premotor cortex exerts both facilitatory and inhibitory control over primary motor cortex during action reprogramming. J Neurosci. 2010 Jan 27;30(4):1395-401. doi: 10.1523/JNEUROSCI.4882-09.2010. PMID 20107065
- [Background] Neubert FX, Mars RB, Buch ER, Olivier E, Rushworth MF. Cortical and subcortical interactions during action reprogramming and their related white matter pathways. Proc Natl Acad Sci U S A. 2010 Jul 27;107(30):13240-5. doi: 10.1073/pnas.1000674107. Epub 2010 Jul 9. PMID 20622155
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552